CLINICAL TRIAL: NCT03167957
Title: A Single-Center, Open-Label, Pilot Study to Evaluate the Efficacy and Safety of Oral Encochleated Amphotericin B (CAMB) in the Treatment of Fluconazole-Resistant Vulvovaginal Candidiasis
Brief Title: Efficacy and Safety of Oral Encochleated Amphotericin B (CAMB) in the Treatment of Fluconazole-Resistant Vulvovaginal Candidiasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer target indication
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB-70008
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Vulvovaginal Candidiases; Yeast Infection; Vulvovaginitis; Yeast Infection Vaginal; Candidiasis, Vulvovaginal
Keywords: fluconazole; fluconazole-resistant
MeSH Terms: conditions — Vulvovaginitis; Candidiasis, Vulvovaginal

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAMB 200 mg (Experimental): 200 mg CAMB Oral Amphotericin B
  Interventions: Drug: Oral Encochleated Amphotericin B (CAMB)
- CAMB 400 mg (Experimental): 400 mg CAMB Oral Amphotericin B
  Interventions: Drug: Oral Encochleated Amphotericin B (CAMB)

INTERVENTIONS:
Drug: Oral Encochleated Amphotericin B (CAMB) — Lipid-crystal nano-particle formulation amphotericin B
  Other Names: MAT2203
  Arms: CAMB 200 mg
Drug: Oral Encochleated Amphotericin B (CAMB) — Lipid-crystal nano-particle formulation amphotericin B
  Other Names: MAT2203
  Arms: CAMB 400 mg

SUMMARY:
This is a single-center, open-label, pilot study to evaluate the efficacy of 14 days of CAMB dosing in subjects with fluconazole-resistant vulvovaginal candidiasis (VVC).

DETAILED DESCRIPTION:
This is a single-center, open-label, pilot study to evaluate the efficacy of 14 days of CAMB dosing in subjects with fluconazole-resistant vulvovaginal candidiasis (VVC).

Approximately 16 women with fluconazole-resistant VVC will be randomized to either 200 mg or 400 mg oral CAMB for 14 days. The primary objectives of this study are to assess the clinical cure rate, mycology eradication and responder outcome. The secondary objective of this study is to evaluate the safety of 200 mg and 400 mg doses of oral CAMB.

ELIGIBILITY:
Inclusion Criteria:

* Female 18-65 years
* Informed Consent
* Clinical diagnosis of fluconazole-resistant VVC
* Negative pregnancy test
* Vaginal pH ≤ 4.5

Exclusion Criteria:

* Intolerance or hypersensitivity to any amphotericin B (AMB) product or to azole antifungal drugs
* Receiving antifungal therapy unrelated to VVC or has evidence of systemic fungal infections requiring antifungal therapy
* Received antifungal treatment for VVC within past 10 days except fluconazole, subjects must discontinue fluconazole after informed consent
* Has another cause or suspected cause of vulvovaginitis
* Has active HPV
* Has other urogenital infection
* Has other vaginal or vulvar condition that would confound interpretation of clinical response
* Has significant laboratory abnormality at screening
* Has Type I diabetes, use of insulin, HbA1c>10
* Exposure to any investigational product within 30 days of screening
* Has other condition that would interfere with subject ability to provide informed consent or put subject at undue risk

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with clinical cure at the Test of Cure visit | 28 days
  Resolution of the VVC signs and symptoms that were present at baseline without further antifungal treatment
The proportion of subjects with mycological eradication at the Test of Cure visit | 28 days
  Negative culture for growth of baseline Candida

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events | 28 days
  Safety assessments include laboratory assessments, vital signs and physical exam

CONTACTS AND LOCATIONS:
Locations (1):
- Tolan Park Clinic, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No